CLINICAL TRIAL: NCT05403229
Title: The Role of Migraine Prophylaxis Agent Topiramate in Treating Patients With Sudden Sensorineural Hearing Loss
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202200324A3C601
Record Dates: First submitted 2022-05-20; First posted 2022-06-03 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Sudden Deafness; Sudden Sensorineural Hearing Loss
Keywords: sudden deafness; SSNHL; migraine; topiramate; sudden sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sudden; Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topiramate arm (Experimental): The experimental group receives a systemic steroid with/without intratympanic steroids as the standard treatment of SSNHL.
  The experimental group receives additional oral topiramate for 6 weeks. The dosage of topiramate is 25 mg orally before bedtime with the weekly escalation of 25 mg up to 100 mg. The total duration of oral topiramate is 6 weeks.
  Interventions: Drug: Topiramate; Drug: Systemic Steroids
- Control arm (Active Comparator): The control arm receives a systemic steroid with/without intratympanic steroids as the standard treatment of SSNHL.
  Interventions: Drug: Systemic Steroids

INTERVENTIONS:
Drug: Topiramate — The topiramate arm receives additional oral topiramate for 6 weeks. The dose of topiramate is started from 25mg orally daily with the weekly escalation of 25mg to a maximum of 100mg.
  Arms: Topiramate arm
Drug: Systemic Steroids — Both groups receive a systemic steroid with/without intratympanic steroids as the standard treatment of SSNHL.

SUMMARY:
Migraine and sudden sensorineural hearing loss(SSNHL) are two related disorders. A systemic steroid is usually used to treat SSNHL but the role of migraine prophylaxis medication remained unknown. Mehdi Abouzari et al. found a better improvement when combining topiramate and nortriptyline with steroids in a retrospective study. However, a prospective study with randomization is needed to elucidate the efficacy of these agents.

This is a clinical study using medication approved and currently prescribed in the clinic. The included patients were those who came to the clinic and were diagnosed with SSNHL within 14 days of onset. Those patients were asked whether they agreed to participate in this clinical trial. Patients who were diagnosed with SSNHL but were later found to be other diseases such as Meniere's disease and cerebellopontine angle will be excluded from this study.

The involved patients were randomized divided into two groups. Both groups received systemic steroids with/without intratympanic steroids. The experimental group receives additional oral topiramate for 6 weeks.

Follow-up time is at least 3 months.

This study is multi-center. Location of the study is performed at Chang gung memorial hospital Linkou branch, Taipei branch, Taoyuan branch, and New Taipei Municipal Tucheng Hospital.

DETAILED DESCRIPTION:
Once the patients were diagnosed with SSNHL, detailed information of the clinical trial will be introduced. If the patient agreed to participate, he/she will be randomized. The experimental group receives additional oral topiramate for 6 weeks.

Both groups follow up at the clinic for at least 3 months. The pure tone audiometry and speech audiometry will be measured at the initial and end of follow-up.

Patients who were later diagnosed with cerebellopontine angle tumors, stroke, or Meniere's disease, will be excluded from this study.

The audiometry and other hearing outcomes will be analyzed at the end of the study. The treatment efficacy, and prognostic factors will be analyzed and reported. Data regarding adverse effects and drop-out will also be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20
* Confirmed diagnosis of unilateral sudden sensorineural hearing loss(SSNHL)
* Treatment started 14 days within onset of SSNHL

Exclusion Criteria:

* Previous SSNHL history
* Previous middle ear disorder such as chronic otitis media, or previous ear surgery
* Meniere's disease and fluctuating hearing loss patients
* Pregnancy or trying to become pregnant
* Leukemia, hemodialysis, and patients who received chemotherapy before.
* Previous head and neck radiotherapy
* cerebellopontine angle tumors such as vestibular schwannoma
* Patients with moderate to severe hepatic insufficiency
* Patients with major depression disorder or suicide attempt
* Patients with glaucoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Audiometry change | Baseline pure tone audiometry will be measured at the time of recruitment. The audiometry will be followed up 3 months after the initial recruitment. The audiometry change between two arms will be calculated and analyzed at the study completion.
  The improvement rate and gain of pure tone audiometry (compare day 0 and day 84)

SECONDARY OUTCOMES:
Audiometry change | The word recognition score will be measured at the time of recruitment(day 0) and end of study(day 84). The pure tone audiometry will be measured at day 56 and improvement would be calculated.
  The improvement rate and gain of word recognition score (compare day 0 and day 84). The improvement rate and gain of pure tone audiometry (compare day 0 and day 56)

CONTACTS AND LOCATIONS:
Overall Officials: BANG-YAN ZHANG, MD., Study Chair — New Taipei Municipal TuCheng Hospital (Built and Operated by Chang Gung Medical Foundation)
Locations (1):
- New Taipei Municipal Tucheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared under the regulation of the institution review board of Chang Gung medical foundation.

REFERENCES:
- [Background] Abouzari M, Goshtasbi K, Chua JT, Tan D, Sarna B, Saber T, Lin HW, Djalilian HR. Adjuvant Migraine Medications in the Treatment of Sudden Sensorineural Hearing Loss. Laryngoscope. 2021 Jan;131(1):E283-E288. doi: 10.1002/lary.28618. Epub 2020 Apr 3. PMID 32243585

DOCUMENTS (1):
  • Study Protocol (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT05403229/Prot_000.pdf